CLINICAL TRIAL: NCT01045330
Title: Effect of the National Taiwan University Hospital Elder Life Program
Brief Title: a Modified NTU-HELP Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other); National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 200803077R
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2013-05

CONDITIONS: Early Ambulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care Group (No Intervention): Usual care consists of standard hospital services provided by physicians, nurses, and support staff (e.g., physical therapist, dietitian) in the general surgery units.
- Experimental Group (Experimental): The intervention consisted of a daily inpatient care protocol on three core intervention protocols on top of hospital routine care.
  Interventions: Behavioral: a modified NTU-HELP

INTERVENTIONS:
Behavioral: a modified NTU-HELP — The intervention consists of a daily inpatient care protocol on three core intervention protocols on top of hospital routine care.
  Arms: Experimental Group

SUMMARY:
The aim is to replicate, develop, and pilot test a model of care for the prevention and management of functional decline of older patients during hospitalization.

DETAILED DESCRIPTION:
to develop an intervention protocol that achieves clinical development objectives in a scientifically rigorous and time efficient manner.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 year and older
* Length of Stay is over 6 days
* Able to communicate verbally or in writing

Exclusion Criteria:

* Coma
* Mechanism ventilation
* Aphasia, if communication ability is severely impaired
* Terminal condition with comfort care only, death imminent
* Combative or dangerous behavior
* Severe psychotic disorder that prevents patient from participating in interventions
* Severe dementia (e.g. unable to communicate; MMSE=0). For patients with severe impairment (e.g. MMSE<10), decision to enroll will be made on a case-by-case basis depending on their ability to participate in intervention.
* Respiratory isolation (e.g. tuberculosis). Patients on contact isolation (e.g. vancomycin-resistant enterococcus) or droplet precautions will be enrolled.
* Discharge firmly anticipated within 6 days of admission. Enroll if discharge date unsure
* Refusal by patient or family member.
* Others. Reason to be well documented.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 377 (Actual)
Dates: Start 2009-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Functional status:Barthel Index. | through study completion, an average of 3 months
  Changes from Baseline Barthel Index (BI) scores at 6 weeks after discharge
Mini-Nutritional Assessment scores (MNA) | through study completion, an average of 3 months
  Changes from Baseline Mini-Nutritional Assessment (MNA) scores at 6 weeks after discharge
Mini Mental State Examination scores (MMSE) | through study completion, an average of 3 months
  Changes from Baseline Mini Mental State Examination (MMSE) scores at 6 weeks after discharge
Frailty rates and transition between frailty states | through study completion, an average of 3 months
  Changes from Baseline Frailty rates at 6 weeks after discharge
Postoperative delirium incidence rate [Confusion Assessment Method (CAM)] | through study completion, an average of 3 months
  Record the incidence of postoperative delirium developing during hospitalization after surgery
Postoperative bowel dysmotility | through study completion, an average of 3 months
  Record the incidence of postoperative bowel dysmotility developing during hospitalization after surgery

SECONDARY OUTCOMES:
Body weight | through study completion, an average of 3 months
  Changes from Baseline Body weight at 6 weeks after discharge
Grip strength | through study completion, an average of 3 months
  Changes from Baseline Grip strength at 6 weeks after discharge
Oral health | through study completion, an average of 3 months
  i.e., plaque index, screens of swallowing function
Executive function | through study completion, an average of 3 months
  ie.e, color trail test
Geriatric Depressive Scale scores (GDS) | through study completion, an average of 3 months
  Changes from Baseline Geriatric Depressive Scale scores (GDS) at 6 weeks after discharge
Length of Hospital Stay (LOS) | through study completion, an average of 3 months
  Record the length of hospital stay for abdominal surgery

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Chai-Hui Chen, DNSc, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan Unversity Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chen CC, Li HC, Liang JT, Lai IR, Purnomo JDT, Yang YT, Lin BR, Huang J, Yang CY, Tien YW, Chen CN, Lin MT, Huang GH, Inouye SK. Effect of a Modified Hospital Elder Life Program on Delirium and Length of Hospital Stay in Patients Undergoing Abdominal Surgery: A Cluster Randomized Clinical Trial. JAMA Surg. 2017 Sep 1;152(9):827-834. doi: 10.1001/jamasurg.2017.1083. PMID 28538964

DOCUMENTS (1):
  • Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT01045330/SAP_000.pdf